CLINICAL TRIAL: NCT04071717
Title: Real-time Neurofeedback Regulating Brain Cognitive Function in Obese Individuals: a Near-infrared Spectroscopy-based Study.
Brief Title: Real-time NIRS Neurofeedback Regulating Brain Cognitive Function in Obese Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wu Wenjun-1 (Other)
Collaborators: Xidian University (Other)
Responsible Party: Sponsor-Investigator, Wu Wenjun-1, Clinical physician, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20192043-F-1
Record Dates: First submitted 2019-07-26; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Neurofeedback
Keywords: NIRS; fNIRS; Neurofeedback; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NIRS group (Experimental): Participants with obesity, 12 sessions of NIRS feedback
  Interventions: Behavioral: NIRS neurofeedback
- Sham NIRS group (Sham Comparator): Participants with obesity, 12 sessions of sham NIRS feedback
  Interventions: Behavioral: Sham NIRS neurofeedback
- Healthy control group (Other): Healthy participants, 12 sessions of NIRS feedback
  Interventions: Behavioral: NIRS neurofeedback

INTERVENTIONS:
Behavioral: NIRS neurofeedback — Neurofeedback as a treatment for people which can be interpreted as a way to increase behavioral inhibition. A method to assess brain activity is functional near-infrared spectroscopy (NIRS), measuring hemodynamic correlates of neural activity.
  Arms: Healthy control group; NIRS group
Behavioral: Sham NIRS neurofeedback — Sham NIRS neurofeedback
  Arms: Sham NIRS group

SUMMARY:
To determine the efficacy of real-time fNIRS neurofeedback for regulating the brain cognitive function in obese individuals.

DETAILED DESCRIPTION:
In the current study, 60 obese subjects will be recruited, and they were randomly classified into the group who will receive real neurofeedback and the group who will receive sham neurofeedback. Participants will receive the real-time neurofeedback for 12 times, 3 to 4 times a week, each time the real-time neurofeedback consists of 12 sessions of liftstone as the index reflecting the brain activity. Sham group will receive the identical neurofeedback.

All of the subjects will undergo magnetic resonance imaging scan, during which T1, diffusion tensor imaging, resting-state, and task fMRI data will be collected. For task Fmri scan, the participants will be asked to finish four cognitive task, including 2-Back working memory, Go/No-Go task, Willingness to Pay for Food, and Delay Discounting tasks. Clinical measurements including BMI, eating behavior, psychiatric status will be assessed. Those aforementioned examinations will be performed at before the neurofeedback, 6th times and the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥ 25
2. 18 to 65 years old
3. No severe mental disorders(depression; schizophrenia; bipolar disorder; etc.).

Exclusion Criteria:

1. Severe dysfunction of heart, liver, kidney and hematopoietic system
2. Substance addiction
3. Patients who cannot be treated with fMRI or fNRIS neurofeedback
4. Those who take other weight loss drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Body Mass Index | Baseline, through study completion, an average of 6 weeks
  Change of the degree of obesity and health of the body

SECONDARY OUTCOMES:
Change of Result of Willingness to Pay for Food | Baseline, through study completion, an average of 6 weeks
  The Willingness to Pay for Food (WTP) task is designed to evaluate obese subjects' cognitive decision ability regarding food. Participants are provided with four response options (i.e. 5¥，30¥，70¥，100¥) that can be selected to purchase a series of visually presented food items (HC, High-calorie food and LC, Low-calorie food).The task will record subjects' response time (RT) and money values selected for each presented food items. Mean response time and mean money values selected for HC food and LC food will be calculated and reported respectively. Shorter RT and bigger more money values selected for LC food represents better outcome. Shorter RT and bigger more money values selected for HC food represents worse outcome.
Change of Result of Go/No-Go | Baseline, through study completion, an average of 6 weeks
  The Go/No-Go task is designed to evaluate subjects' inhibitory control capacity.
  Participants were instructed to press a button as quickly and accurately as possible in response to go trials and to refrain from responding to no-go trials. The current task involved two conditions (Go-condition and NoGo-condition). The task will record subjects' response time (RT) and whether correct for each trial response. Task response accuracy, response time, omission error rate (OE, %) and commission error rate (CE, %) will be calculated and reported. Omission error rate (OE, %) was calculated by dividing the total number of non-responses to go-items by the total number of go-trials. Commission error rate (CE, %) was calculated by dividing the total number of incorrect responses to no-go trials by the total number of no-go trials. Higher accuracy, lower RT, lower OE and lower CE represent better treatment outcome.
Working Memory | Baseline, through study completion, an average of 6 weeks
  The Working Memory task (WM) is designed to evaluate obese subjects' short-term memory. Subjects performed food pictures variant version of working memory (n-back) tasks, which were block designed. In 0-back blocks (including 0-back block for HC (High-calorie food), LC (Low-calorie food) and Neutral pictures respectively), subjects were required to identify a single prespecified picture. Briefly, subjects were asked to press a button as quickly to indicate whether a picture presented on a screen matched the picture previously presented.The task will record subjects' response time (RT) and accuracy for each n-back block. Subjects' 2-back response time and accuracy for HC and LC will be calculated and reported. Shorter RT and higher accuracy of 2-back for HC and LC represents better outcome. Longer RT and lower accuracy of 2-back for HC and LC represents worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjun Wu, Master, Study Chair — Xijing Hospital, The Air Force Medical University; Huaning Wang, Doctor, Principal Investigator — Xijing Hospital, The Air Force Medical University; Yi Zhang, professor, Principal Investigator — Xidian University
Locations (1):
- Department of Psychiatry, Xijing Hospital, The Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Samuel I, Mason EE, Renquist KE, Huang YH, Zimmerman MB, Jamal M. Bariatric surgery trends: an 18-year report from the International Bariatric Surgery Registry. Am J Surg. 2006 Nov;192(5):657-62. doi: 10.1016/j.amjsurg.2006.07.006. PMID 17071202
- [Result] Watanabe T, Sasaki Y, Shibata K, Kawato M. Advances in fMRI Real-Time Neurofeedback: (Trends in Cognitive Sciences 21, 997-1010, 2017). Trends Cogn Sci. 2018 Aug;22(8):738. doi: 10.1016/j.tics.2018.05.007. Epub 2018 Jun 1. No abstract available. PMID 29866489
- [Result] Schwartz DH, Leonard G, Perron M, Richer L, Syme C, Veillette S, Pausova Z, Paus T. Visceral fat is associated with lower executive functioning in adolescents. Int J Obes (Lond). 2013 Oct;37(10):1336-43. doi: 10.1038/ijo.2013.104. Epub 2013 Jun 5. PMID 23797144
- [Result] Diamantis T, Apostolou KG, Alexandrou A, Griniatsos J, Felekouras E, Tsigris C. Review of long-term weight loss results after laparoscopic sleeve gastrectomy. Surg Obes Relat Dis. 2014 Jan-Feb;10(1):177-83. doi: 10.1016/j.soard.2013.11.007. Epub 2013 Nov 21. PMID 24507083